CLINICAL TRIAL: NCT07325448
Title: Assessing MB-Spirit: A Novel Intervention for Promoting Spiritual Development and Psychological Well-being
Brief Title: Assessing MB-Spirit for Psychological Well-being
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sara W Lazar (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Sponsor-Investigator, Sara W Lazar, Associate Research Scientist, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025A014112
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Stress
Keywords: stress; MRI; spirituality; well-being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MB-Spirit (Experimental): 8-week online course that combines mindfulness with character strengths to promote well-being
  Interventions: Behavioral: MB-Spirit
- Wait-list (No Intervention): Wait list

INTERVENTIONS:
Behavioral: MB-Spirit — 8-week online course that uses character strengths and mindfulness to promote well-being. Based on 3-part model of spirituality
  Arms: MB-Spirit

SUMMARY:
The goal of this clinical trial is to learn if a new behavioral intervention, MB-Spirit, can improve well-being in stressed adults. The main questions it aims to answer are:

1. Can MB-Spirit improve well-being?
2. What brain changes accompany participation in MB-Spirit?

Participants will:

1. Be enrolled in an online course that meets for two hours every week for 8-weeks.
2. Complete questionnaires before and after the course.
3. Complete an MRI scan of their brain before and after the course.

Participants will be randomized to either take the course right away, or be put on a wait-list. Those on the wait-list will undergo the testing at 2 timepoints before they start the program.

DETAILED DESCRIPTION:
Forty-four individuals with high stress will be randomized 1:1, stratified by sex, to either MB-SPIRIT or wait-list. Participants will receive daily email with a link to a REDCap database to record minutes of formal meditation practice. Pre and post testing will occur within a 21-day testing period before or after the intervention. We will assess changes in spiritual well-being (Primary outcome), mindfulness, and use of character/virtue strengths (secondary outcomes). Changes in clinical symptoms will be explored. Participants will also complete a structured interview to assess developmental stage at the baseline time-point. Participants randomized to MB-Spirit will also undergo functional magnetic resonance imaging (fMRI) scanning before and after their program. Scans consist of a high-resolution gray matter scan, a 10-minute resting state scan and three 10-minute guided meditation scans. Participants will rate the 'depth' of each spiritual state they experience while they are in the scanner on a 5-point scale. As a manipulation check, after exiting the scanner they will be asked to describe the non-dual states and which virtues arose. We will also assess the acceptability of the task.

ELIGIBILITY:
Inclusion Criteria:

* Understands English
* Able to attend all 8 classes
* Able to travel to Boston for MRI scans

Exclusion Criteria:

* claustrophobia, pregnancy, head trauma, metallic implants or devices contraindicating MRI, left-handed, conditions that alter cerebral blood flow or metabolism (e.g. stroke), current use of psychotropic medications, lifetime history of suicidality, homicidally, self-destructive acts, schizophrenia or psychosis.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
FACIT-SP meaning and peace subscale | 8 weeks
  The meaning and peace subscale of the widely used and well-validated FACIT-SP-non-illness (Functional assessment of chronic illness therapy spiritual wellbeing - non illness) is our primary outcome metric. It has very good reliability (alpha=.81) and has high discriminate validity.

SECONDARY OUTCOMES:
Duke University Religion Index | 8-weeks
  Duke University Religion Index (DUREL) is a five-item measure to assess religiosity by examining three key dimensions: organizational religious activity (e.g., attending services), non-organizational religious activity (e.g., private prayer), and intrinsic religiosity (e.g., personal religious commitment and its influence on life). The overall scale has high test-retest reliability (intra-class correlation = 0.91), high internal consistence (Cronbach's alpha's = 0.78-0.91), high convergent validity with other measures of religiosity (r's = 0.71-0.86).
Brief Signature Strengths Use Scale (BSSUS) | 8 weeks
  Brief Signature Strengths Use Scale (BSSUS) measures the extent to which participants recognize and use their signature character strengths. Five items are scored on a 7-point Likert scale, ranging from ranging from Strongly disagree to Very strongly agree. Higher scores indicate higher strength use.
Metacognitive Processes of Decentering Scale (MPoD-t) | 8 weeks
  The Metacognitive Processes of Decentering Scale (MPoD-t) is a self-report scale developed to measure the ability to decenter, or separate one's sense of self from internal experiences, by assessing three core metacognitive processes: meta-awareness, (dis)identification with internal states, and (non)reactivity to thought content. The MPoD-t scales are used to study decentering, its role in mental health, and its potential as a therapeutic mechanism in mindfulness-based interventions
PROMIS-29 | 8 weeks
  The 29-item PROMIS-29 contains short assessments of eight core health domains including: anxiety, depression, physical function, sleep disturbance, pain interference and pain intensity, fatigue, and ability to participate in social roles and activities. Cronbach's α reliability for all domains range from 0.77 to 0.98 and scores remained stable over 18 months132 All domains use a 7-day recall period, except for PF and SRAA.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Lazar, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Charlestown Navy Yard Campus, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified data will be shared with other researchers. We are collaborating with an investigator at the University of Vienna who will have access to all de-identified data.
Time Frame: The brain and self-report data and meta-data will be deposited in the ENIGMA-Meditation data repository hosted at Ohio State University within 6 months of the first paper being accepted for publication. There are no plans to remove the data from the repository.
Access Criteria: No identifiable information will be included in the dataset. Any researcher interested in accessing the data must first contact the study PI and request permission. The study PI then needs to obtain IRB approval for any additional analyses that will be performed.